CLINICAL TRIAL: NCT00257699
Title: Metronidazole and Ciprofloxacin in the Treatment of Colonic Crohn's Disease: The MACINTOCC Trial.
Brief Title: Study of Antibiotics in the Treatment of Colonic Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate recruitment to meet completion date
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSH REB 04-0257-A
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Randomized; Ciprofloxacin; Metronidazole; Antibiotic
MeSH Terms: conditions — Crohn Disease | interventions — Ciprofloxacin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- I (Placebo Comparator): Ciprofloxacin placebo and Metronidazole placebo
  Interventions: Drug: Metronidazole placebo; Drug: ciprofloxacin placebo
- II (Experimental): Ciprofloxacin 500 mg bid po Metronidazole - total daily dose dependent on body weight
  Interventions: Drug: ciprofloxacin; Drug: metronidazole

INTERVENTIONS:
Drug: Metronidazole placebo
  Arms: I
Drug: ciprofloxacin placebo
  Arms: I
Drug: ciprofloxacin — 500 mg bid po
  Other Names: Cipro
  Arms: II
Drug: metronidazole — 250 mg bid po / 250 mg tid po / 500 mg bid po depending on body weight
  Other Names: Flagyl
  Arms: II

SUMMARY:
Crohn's disease (CD) is a form of inflammatory bowel disease that can affect any part of the digestive system. Symptoms of this chronic illness include abdominal pain, bloating, nausea, vomiting, and diarrhea. CD also causes bowel wall ulcers, strictures (narrowings of a hollow structure due to scar tissue and swelling), and fistulae (abnormal passages from the intestines to another organ or to the skin).

CD is thought to arise from a combination of inherited (genetic) factors and some undefined environmental factor(s). One environmental factor that has been shown to be intimately involved with the development of CD is the presence of bacteria that normally inhabit the intestines. As a result, some physicians have tried to alter the normal bacterial population as a means of controlling the inflammation (swelling) in the intestines of individuals with CD. Among such strategies is the use of a combination of metronidazole and ciprofloxacin. These broad-spectrum antibiotics control CD symptoms by acting on the intestinal bacteria that can contribute to chronic inflammation. More investigation is needed to firmly establish the usefulness of this therapy because previous clinical trials have given mixed results, although they have suggested that antibiotics can be particularly useful in cases of Crohn's colitis (CD that primarily affects the large intestine). Because these earlier studies have lacked a large enough patient population with colonic involvement, a trial focusing on this CD subgroup with a sufficient number of subjects will help to clarify the value of combining metronidazole and ciprofloxacin.

The proposed study will test the hypothesis that combination antibiotic therapy is effective in the treatment of CD involving the colon. The study will compare the use of combination therapy consisting of metronidazole and ciprofloxacin with placebo (dummy tablets) and will examine the results of treatment at the end of 8 weeks of treatment.

DETAILED DESCRIPTION:
The role of bacteria and microbial agents in the pathogenesis of Crohn's disease has been suggested and is supported by animal models of inflammatory bowel disease (IBD) in which the presence of normal gut flora is required for the initiation and full expression of the inflammatory reaction. In human Crohn's disease, antibiotics are commonly used even though the evidence to support this practice is not strong. Several studies have indicated that antibiotics have some biological activity in Crohn's disease and that this activity may be most pronounced in the subset of patients with colonic involvement.

In order to better justify the use of antibiotics in the treatment of Crohn's disease, the Antibiotics for Colonic Crohn's Disease trial has been designed to determine if ciprofloxacin and metronidazole combination therapy is effective in the treatment of active Crohn's disease of the colon. This two arm, multi-centre, randomized, double-blind, parallel-group, placebo-controlled study will involve 136 patients with mild to moderate active Crohn's disease of the colon (with or without ileal involvement), as defined by a Crohn's Disease Activity Index (CDAI) score between 220 and 450.

Eligible patients will be randomly assigned to receive one of two treatment regimens: (1) ciprofloxacin (500 mg po bid; provided as

1 x 500 mg tablets) and metronidazole (<50 kg, 250 mg po bid; 50-75 kg, 250 mg po tid; >75 kg, 500 mg po bid; all doses provided as 1 x 250 mg tablets) or (2) placebo. Treatment will be continued for a period of 8 weeks.

Treatment success will be defined as a complete response to therapy at the end of eight weeks. Complete response (remission) will be defined as a reduction of the CDAI score to below 150 points with a reduction of at least 70 points from baseline. Partial response (improvement) will be analyzed as a secondary outcome measure and will be defined as a reduction of the CDAI score by 70 points or more but with a final value of 150 points or greater. Patients who experience a persistent rise in their CDAI scores of 100 points or more on two consecutive visits or a rise in their CDAI score to 400 points or more at any visit will be considered to be treatment failures and will be withdrawn from the study.

The primary analysis will be an intent-to-treat comparison of the proportion of patients achieving remission by 8 weeks in the ciprofloxacin/metronidazole and placebo groups. Secondary outcome measures will evaluate partial response and adverse event rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 16 years of age or older.
* Patients who have been diagnosed with Crohn's disease for more than 1 month.
* Patients with CDAI scores between 220 and 450 at the randomization visit.
* Patients with Crohn's disease involving any portion of the colon (more than erythema and/or 10 aphthoid ulcers) with or without distal or terminal ileal disease. (Subjects may have had previous partial colonic resection consisting of less than 50% of the estimated length of the colon.)

Exclusion Criteria:

* Female patients who are, or may become, pregnant during the course of the study or women who are breastfeeding.
* Patients who have an allergy or contraindication to ciprofloxacin or to metronidazole.
* Patients who are experiencing a complication of Crohn's disease (e.g. perforation, acute obstruction, hemorrhage) requiring urgent surgical intervention.
* Patients with subacute small bowel obstruction.
* Patients with significant, symptomatic Crohn's disease of the esophagus, the stomach, the duodenum, or the jejunum.
* Patients who have received, i)any antibiotic within 2 weeks of the screening visit, ii)systemic corticosteroid therapy within 2 weeks of the screening visit, iii)parenteral nutritional therapy within 2 weeks of the screening visit, iv)enteral elemental or polymeric nutritional therapy or exclusively liquid diet within 2 weeks of the screening visit, v) infliximab within 12 weeks of the screening visit, vi)an initiation of therapy with sulphasalazine or with any 5-ASA preparation within 4 weeks of the screening visit or a change in the dose within 2 weeks of the screening visit (Patients on stable doses of sulphasalazine or of a 5-ASA preparation for at least 2 weeks prior to the screening visit are eligible for entry into the study if the total duration of the therapy is at least 4 weeks prior to screening.), vii)an initiation of azathioprine, 6-MP, or methotrexate within 12 weeks of the screening visit or changes in the dose of azathioprine, of 6-MP, or of methotrexate within 4 weeks of screening visit (Patients receiving azathioprine, 6-MP, or methotrexate for at least 12 weeks and at a stable dose for at least 4 weeks prior to the screening visit are eligible for inclusion.), viii)other therapy not listed above for Crohn's disease within 4 weeks of the screening visit, AND/OR ix)any investigational drug within 12 weeks of the screening visit.
* Patients whose stool culture tests positive for enteric pathogens at the screening visit.
* Patients whose stool assay is positive for Clostridium difficile toxin at the screening visit.
* Patients who have another clinically significant medical or psychiatric illness (as judged by the investigator).
* Patients who have had a resection of more than 100 cm of their small intestine, more than half of their colon, or who have an ileostomy.
* Patients who are unable to provide informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Complete response to therapy defined as a reduction of the CDAI score to below 150 points with a reduction of at least 70 points from baseline. | 8 weeks

SECONDARY OUTCOMES:
Partial response (improvement) will be analyzed as a secondary outcome measure and will be defined as a reduction of the CDAI score by 70 points or more but with a final value of 150 points or greater. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: A. Hillary Steinhart, M.D., Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada